CLINICAL TRIAL: NCT01813695
Title: Preemptive Genotyping of Children and Adolescents at Risk for Surgery and Subsequent Pain Management
Brief Title: Preemptive Genotyping and Pain Management
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-0853; NIH 3U01 HG006828-01S1 (Other Grant/Funding Number: NIH Supplement Award)
Record Dates: First submitted 2013-03-11; First posted 2013-03-19 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Pain
Keywords: Preemptive genetic testing; Pain; Pediatrics; Orthopedics; Pectus excavatum; Scoliosis
MeSH Terms: conditions — Pain; Funnel Chest; Scoliosis | interventions — Medical Records; Electronic Health Records

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preemptive: Patients with genotype testing entered into electronic medical record for consideration and opioid administration postoperatively.
  Interventions: Procedure: Preemptive genotyping in medical record
- Control: Genetic sample taken but withheld from electronic medical record.
  Interventions: Procedure: Genotyping not included in electronic medical record

INTERVENTIONS:
Procedure: Preemptive genotyping in medical record
  Groups: Preemptive
Procedure: Genotyping not included in electronic medical record
  Groups: Control

SUMMARY:
The purpose of this study is to see if testing for genes related to pain and pain management before surgery affects how patients are treated for pain after surgery. The investigators want to know if this information will be used to effectively treat patients for pain after surgery if the clinical staff have a chance to review it before the surgery.

DETAILED DESCRIPTION:
Purpose: To determine the feasibility of preemptive (preoperative) cytochrome P450 isoenzyme (CYP2D6) testing and the variability of clinical measures (postoperative) in children whose opioid selection and dosing is influenced by preemptive CYP2D6 testing compared to children whose pain management does not include CYP2D6 preemptive testing. Results from this pilot study will inform a future study investigating the utility of preemptive pharmacogenomic testing in children at risk for requiring inpatient acute pain management with opioids.

ELIGIBILITY:
Inclusion Criteria:

* Children, 6-17 years of age and adults, 18 - 21 years with idiopathic scoliosis and/or pectus excavatum scheduled for surgical clinic visit
* BMI < 30
* Cognitively able to use a 0 - 10 numerical rating scale (NRS) to report level of pain
* Parents give permission (and children give assent when appropriate) or adult participants give consent for CYP2D6 results to be placed in Cincinnati Children's Hospital Medical Center (CCHMC's) EPIC

Exclusion Criteria:

* • Who had prior surgery for idiopathic scoliosis and/or pectus excavatum

  * Who have prior CYP2D6 testing or Genetic Pharmacology Service (GPS) Psychiatry Panel documented in EPIC
  * Who are taking prescription medication known to inhibit or induce CYP2D6
  * Who are taking prescription medication known to inhibit (e.g. voriconazole) or induce (e.g. carbamazepine and rifampin) CYP3A4
  * Who have liver or renal failure
  * Who have history of narcotic abuse

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients scheduled for scoliosis and pectus excavatum surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2013-03; Primary Completion 2020-11-04 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of PreEmptive Genotyping Testing | From initial clinic visit to post-operative discharge, expected average of three months
  The Investigator will use descriptive and summary statistics to determine the feasibility of preemptive CYP2D6 testing in children evaluated during a clinic visit for potential surgery.

SECONDARY OUTCOMES:
Analgesia Effectiveness | Admission for surgery, up to two weeks
  Pain score (NRS 0 - 10) before and after each oral opioid dose (we will use time between the before and after pain score measures as a covariate)
Analgesia Toxicity | Admission for surgery, up to two weeks
  1. At least 1 documented ADR;
  2. Total number of documented ADRs;
  3. Total number of ADR related responses in "Pain Medicine Report" answered "sometimes" or "always";
  4. Total number of documented GI related ADRs - nausea (yes/no) and vomiting (yes/no);
  5. Total number of documented central nervous system (CNS) ADRs (Modified Ramsay scores > 4 and respiratory rate (RR) indicative of respiratory depression; and oxygen saturations (SpO2) < 90% on room air; and need for supplemental oxygen; and response of "always" for "Pain Medicine Report" question, "When you took the pain medicine, how often did it make you fall asleep?"
Analgesia Effectiveness | Admission for surgery, up to two weeks
  Participant related responses in "Pain Medicine Report"
Analgesia Effectiveness | Admission for surgery, up to two weeks
  Total number of rescue IV pain medication doses
Analgesia Effectiveness | Admission for surgery, up to two weeks
  Total number of concomitant analgesic adjunct medications such as muscle relaxants, acetaminophen.
Analgesia Effectiveness | Admission for surgery, up to two weeks
  Total mg/kg 24hr dose of oral opioids

OTHER OUTCOMES:
Association between specific genotypes and pain sensitivity, reported postoperative pain, and opioid response | Postoperative surgery, up to two weeks
  To explore association between specific genotypes (in addition to CYP2D6) and pain sensitivity, reported postoperative pain, and opioid response (pain reduction and incidence of adverse drug reactions (ADRs))

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Sadhasivam, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadhasivam S, Boat A, Mahmoud M. Comparison of patient-controlled analgesia with and without dexmedetomidine following spine surgery in children. J Clin Anesth. 2009 Nov;21(7):493-501. doi: 10.1016/j.jclinane.2008.12.017. PMID 20006257
- [Background] Voepel-Lewis T, Marinkovic A, Kostrzewa A, Tait AR, Malviya S. The prevalence of and risk factors for adverse events in children receiving patient-controlled analgesia by proxy or patient-controlled analgesia after surgery. Anesth Analg. 2008 Jul;107(1):70-5. doi: 10.1213/ane.0b013e318172fa9e. PMID 18635469
- [Background] Aubrun F, Monsel S, Langeron O, Coriat P, Riou B. Postoperative titration of intravenous morphine. Eur J Anaesthesiol. 2001 Mar;18(3):159-65. doi: 10.1046/j.0265-0215.2000.00796.x. PMID 11298174
- [Background] Ross JR, Rutter D, Welsh K, Joel SP, Goller K, Wells AU, Du Bois R, Riley J. Clinical response to morphine in cancer patients and genetic variation in candidate genes. Pharmacogenomics J. 2005;5(5):324-36. doi: 10.1038/sj.tpj.6500327. PMID 16103897
- [Background] D'Arcy Y. One opioid does not fit all. Nurse Pract. 2007 Nov;32(11):7-8. doi: 10.1097/01.NPR.0000298262.47655.14. No abstract available. PMID 18075450
- [Background] Sadhasivam S, Cohen LL, Szabova A, Varughese A, Kurth CD, Willging P, Wang Y, Nick TG, Gunter J. Real-time assessment of perioperative behaviors and prediction of perioperative outcomes. Anesth Analg. 2009 Mar;108(3):822-6. doi: 10.1213/ane.0b013e318195c115. PMID 19224789
- [Background] Beaulieu P, Cyrenne L, Mathews S, Villeneuve E, Vischoff D. Patient-controlled analgesia after spinal fusion for idiopathic scoliosis. Int Orthop. 1996;20(5):295-9. doi: 10.1007/s002640050081. PMID 8930721
- [Background] Dahan A, Aarts L, Smith TW. Incidence, Reversal, and Prevention of Opioid-induced Respiratory Depression. Anesthesiology. 2010 Jan;112(1):226-38. doi: 10.1097/ALN.0b013e3181c38c25. PMID 20010421
- [Background] Hanna MH, Elliott KM, Fung M. Randomized, double-blind study of the analgesic efficacy of morphine-6-glucuronide versus morphine sulfate for postoperative pain in major surgery. Anesthesiology. 2005 Apr;102(4):815-21. doi: 10.1097/00000542-200504000-00018. PMID 15791112
- [Background] Duedahl TH, Hansen EH. A qualitative systematic review of morphine treatment in children with postoperative pain. Paediatr Anaesth. 2007 Aug;17(8):756-74. doi: 10.1111/j.1460-9592.2007.02213.x. PMID 17596221
- [Background] Gramke HF, de Rijke JM, van Kleef M, Raps F, Kessels AG, Peters ML, Sommer M, Marcus MA. The prevalence of postoperative pain in a cross-sectional group of patients after day-case surgery in a university hospital. Clin J Pain. 2007 Jul-Aug;23(6):543-8. doi: 10.1097/AJP.0b013e318074c970. PMID 17575496
- [Background] Sommer M, de Rijke JM, van Kleef M, Kessels AG, Peters ML, Geurts JW, Gramke HF, Marcus MA. The prevalence of postoperative pain in a sample of 1490 surgical inpatients. Eur J Anaesthesiol. 2008 Apr;25(4):267-74. doi: 10.1017/S0265021507003031. Epub 2007 Dec 6. PMID 18053314
- [Background] Fletcher D, Fermanian C, Mardaye A, Aegerter P; Pain and regional anesthesia committee of the French Anesthesia and Intensive Care Society (SFAR). A patient-based national survey on postoperative pain management in France reveals significant achievements and persistent challenges. Pain. 2008 Jul 15;137(2):441-451. doi: 10.1016/j.pain.2008.02.026. Epub 2008 Apr 15. PMID 18417292
- [Background] Brennan F, Carr DB, Cousins M. Pain management: a fundamental human right. Anesth Analg. 2007 Jul;105(1):205-21. doi: 10.1213/01.ane.0000268145.52345.55. PMID 17578977
- [Background] Joshi GP, Kehlet H, Rawal N; PROSPECT Working Group. Evidence-based guidelines for postoperative pain management. Reg Anesth Pain Med. 2007 Mar-Apr;32(2):173. doi: 10.1016/j.rapm.2006.11.002. No abstract available. PMID 17350537
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Raja SN, Jensen TS. Predicting postoperative pain based on preoperative pain perception: are we doing better than the weatherman? Anesthesiology. 2010 Jun;112(6):1311-2. doi: 10.1097/ALN.0b013e3181dcd5cc. No abstract available. PMID 20502114
- [Background] White PF, Kehlet H. Improving postoperative pain management: what are the unresolved issues? Anesthesiology. 2010 Jan;112(1):220-5. doi: 10.1097/ALN.0b013e3181c6316e. No abstract available. PMID 20010418
- [Background] Kim H, Ramsay E, Lee H, Wahl S, Dionne RA. Genome-wide association study of acute post-surgical pain in humans. Pharmacogenomics. 2009 Feb;10(2):171-9. doi: 10.2217/14622416.10.2.171. PMID 19207018
- [Background] Skorpen F, Laugsand EA, Klepstad P, Kaasa S. Variable response to opioid treatment: any genetic predictors within sight? Palliat Med. 2008 Jun;22(4):310-27. doi: 10.1177/0269216308089302. PMID 18541635
- [Background] Kelly LE, Rieder M, van den Anker J, Malkin B, Ross C, Neely MN, Carleton B, Hayden MR, Madadi P, Koren G. More codeine fatalities after tonsillectomy in North American children. Pediatrics. 2012 May;129(5):e1343-7. doi: 10.1542/peds.2011-2538. Epub 2012 Apr 9. PMID 22492761
- [Background] Food and Drug Administration. FDA Drug Safety Communication: Codeine use in certain children after tonsillectomy and/or adenoidectomy may lead to rare, but life-threatening adverse events or death. http://wwwfdagov/Drugs/DrugSafety/ucm313631htm. Accessed 8/15/2012August 15, 2012
- [Background] Shipton EA, Muller FO, Herhold WJ, De Vaal JB. Ingestion of codeine and salicylic acid causing convulsions and coma. A case report. S Afr Med J. 1984 Sep 22;66(12):460. PMID 6484774
- [Background] Kintz P, Tracqui A, Mangin P. Codeine concentrations in human samples in a case of fatal ingestion. Int J Legal Med. 1991;104(3):177-8. doi: 10.1007/BF01369725. PMID 1911418
- [Background] Magnani B, Evans R. Codeine intoxication in the neonate. Pediatrics. 1999 Dec;104(6):e75. doi: 10.1542/peds.104.6.e75. PMID 10586009
- [Background] Voronov P, Przybylo HJ, Jagannathan N. Apnea in a child after oral codeine: a genetic variant - an ultra-rapid metabolizer. Paediatr Anaesth. 2007 Jul;17(7):684-7. doi: 10.1111/j.1460-9592.2006.02182.x. PMID 17564651
- [Background] Ciszkowski C, Madadi P, Phillips MS, Lauwers AE, Koren G. Codeine, ultrarapid-metabolism genotype, and postoperative death. N Engl J Med. 2009 Aug 20;361(8):827-8. doi: 10.1056/NEJMc0904266. No abstract available. PMID 19692698
- [Background] Hermanns-Clausen M, Weinmann W, Auwarter V, Ferreiros N, Trittler R, Muller C, Pahl A, Superti-Furga A, Hentschel R. Drug dosing error with drops: severe clinical course of codeine intoxication in twins. Eur J Pediatr. 2009 Jul;168(7):819-24. doi: 10.1007/s00431-008-0842-7. Epub 2008 Oct 21. PMID 18936971
- [Background] Lalovic B, Phillips B, Risler LL, Howald W, Shen DD. Quantitative contribution of CYP2D6 and CYP3A to oxycodone metabolism in human liver and intestinal microsomes. Drug Metab Dispos. 2004 Apr;32(4):447-54. doi: 10.1124/dmd.32.4.447. PMID 15039299
- [Background] Zwisler ST, Enggaard TP, Mikkelsen S, Brosen K, Sindrup SH. Impact of the CYP2D6 genotype on post-operative intravenous oxycodone analgesia. Acta Anaesthesiol Scand. 2010 Feb;54(2):232-40. doi: 10.1111/j.1399-6576.2009.02104.x. Epub 2009 Aug 31. PMID 19719813
- [Background] Otton SV, Schadel M, Cheung SW, Kaplan HL, Busto UE, Sellers EM. CYP2D6 phenotype determines the metabolic conversion of hydrocodone to hydromorphone. Clin Pharmacol Ther. 1993 Nov;54(5):463-72. doi: 10.1038/clpt.1993.177. PMID 7693389
- [Background] Smith HS. The metabolism of opioid agents and the clinical impact of their active metabolites. Clin J Pain. 2011 Nov-Dec;27(9):824-38. doi: 10.1097/AJP.0b013e31821d8ac1. PMID 21677572
- [Background] Gan SH, Ismail R, Wan Adnan WA, Zulmi W. Impact of CYP2D6 genetic polymorphism on tramadol pharmacokinetics and pharmacodynamics. Mol Diagn Ther. 2007;11(3):171-81. doi: 10.1007/BF03256239. PMID 17570739
- [Background] Andreassen TN, Eftedal I, Klepstad P, Davies A, Bjordal K, Lundstrom S, Kaasa S, Dale O. Do CYP2D6 genotypes reflect oxycodone requirements for cancer patients treated for cancer pain? A cross-sectional multicentre study. Eur J Clin Pharmacol. 2012 Jan;68(1):55-64. doi: 10.1007/s00228-011-1093-5. Epub 2011 Jul 7. PMID 21735164
- [Background] Lam J, Kelly L, Ciszkowski C, Landsmeer ML, Nauta M, Carleton BC, Hayden MR, Madadi P, Koren G. Central nervous system depression of neonates breastfed by mothers receiving oxycodone for postpartum analgesia. J Pediatr. 2012 Jan;160(1):33-7.e2. doi: 10.1016/j.jpeds.2011.06.050. Epub 2011 Aug 31. PMID 21880331
- [Background] Sadhasivam S, Myer CM 3rd. Preventing opioid-related deaths in children undergoing surgery. Pain Med. 2012 Jul;13(7):982-3; author reply 984. doi: 10.1111/j.1526-4637.2012.01419.x. Epub 2012 Jun 13. PMID 22694279
- [Background] Gillen C, Haurand M, Kobelt DJ, Wnendt S. Affinity, potency and efficacy of tramadol and its metabolites at the cloned human mu-opioid receptor. Naunyn Schmiedebergs Arch Pharmacol. 2000 Aug;362(2):116-21. doi: 10.1007/s002100000266. PMID 10961373
- [Background] Stamer UM, Lehnen K, Hothker F, Bayerer B, Wolf S, Hoeft A, Stuber F. Impact of CYP2D6 genotype on postoperative tramadol analgesia. Pain. 2003 Sep;105(1-2):231-8. doi: 10.1016/s0304-3959(03)00212-4. PMID 14499440
- [Background] Crews KR, Gaedigk A, Dunnenberger HM, Klein TE, Shen DD, Callaghan JT, Kharasch ED, Skaar TC; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium (CPIC) guidelines for codeine therapy in the context of cytochrome P450 2D6 (CYP2D6) genotype. Clin Pharmacol Ther. 2012 Feb;91(2):321-6. doi: 10.1038/clpt.2011.287. Epub 2011 Dec 28. PMID 22205192
- [Background] Lovlie R, Daly AK, Molven A, Idle JR, Steen VM. Ultrarapid metabolizers of debrisoquine: characterization and PCR-based detection of alleles with duplication of the CYP2D6 gene. FEBS Lett. 1996 Aug 19;392(1):30-4. doi: 10.1016/0014-5793(96)00779-x. PMID 8769309
- [Background] von Baeyer CL, Spagrud LJ, McCormick JC, Choo E, Neville K, Connelly MA. Three new datasets supporting use of the Numerical Rating Scale (NRS-11) for children's self-reports of pain intensity. Pain. 2009 Jun;143(3):223-227. doi: 10.1016/j.pain.2009.03.002. Epub 2009 Apr 8. PMID 19359097
- [Background] Bulloch B, Tenenbein M. Validation of 2 pain scales for use in the pediatric emergency department. Pediatrics. 2002 Sep;110(3):e33. doi: 10.1542/peds.110.3.e33. PMID 12205283
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Ramsay MA. Anesthesia and pain management at Baylor University Medical Center. Proc (Bayl Univ Med Cent). 2000 Apr;13(2):151-65. doi: 10.1080/08998280.2000.11927660. No abstract available. PMID 16389370
- [Background] Paqueron X, Lumbroso A, Mergoni P, Aubrun F, Langeron O, Coriat P, Riou B. Is morphine-induced sedation synonymous with analgesia during intravenous morphine titration? Br J Anaesth. 2002 Nov;89(5):697-701. PMID 12393765
- [Background] Whitlock MC. Combining probability from independent tests: the weighted Z-method is superior to Fisher's approach. J Evol Biol. 2005 Sep;18(5):1368-73. doi: 10.1111/j.1420-9101.2005.00917.x. PMID 16135132
- [Derived] Packiasabapathy S, Zhang X, Ding L, Aruldhas BW, Pawale D, Sadhasivam S. Quantitative Pupillometry as a Predictor of Pediatric Postoperative Opioid-Induced Respiratory Depression. Anesth Analg. 2021 Oct 1;133(4):991-999. doi: 10.1213/ANE.0000000000005579. PMID 34029273